CLINICAL TRIAL: NCT04087811
Title: Postmarket Registry for Evaluation of the Superion® Spacer
Acronym: PRESS
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-VISS-01
Record Dates: First submitted 2019-06-05; First posted 2019-09-12 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-06

CONDITIONS: Lumbar Spinal Stenosis
Keywords: LSS
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Superion® Indirect Decompression System (IDS): Superion® Indirect Decompression System (IDS) - Interspinous Spacer
  Interventions: Device: Superion® Indirect Decompression System (IDS)

INTERVENTIONS:
Device: Superion® Indirect Decompression System (IDS) — Superion® Indirect Decompression System (IDS) (Superion® implant)

SUMMARY:
To gather evidence documenting the performance and clinical outcomes associated with treatment of moderate degenerative lumbar spinal stenosis using the Superion® Indirect Decompression System (IDS).

DETAILED DESCRIPTION:
To gather evidence documenting the performance and clinical outcomes associated with treatment of moderate degenerative lumbar spinal stenosis using the Superion® IDS in patients ≥45 years of age suffering from symptoms of neurogenic intermittent claudication secondary to a confirmed diagnosis of moderate degenerative lumbar spinal stenosis at one or two contiguous levels from L1 to L5.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients ≥45 years of age
* symptoms of neurogenic intermittent claudication and a confirmed diagnosis of moderate degenerative lumbar stenosis at one or two contiguous levels from L1 to L5
* meeting the labeled indications for use of the Superion® Indirect Decompression System (IDS)

Exclusion Criteria:

* not contraindicated as described in the labeled indications for use

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from symptoms of neurogenic intermittent claudication secondary to a confirmed diagnosis of moderate degenerative lumbar spinal stenosis
Sampling Method: Non-Probability Sample
Enrollment: 1674 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (66):
- United States (66):
  - (ACT) Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - HOPE Research Institute, Scottsdale, Arizona
  - NuVation Pain Group, Buena Park, California
  - Comprehensive Pain Physicians, Burbank, California
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - Pain Medicine Associates, Fountain Valley, California
  - Valley Pain Management, Fresno, California
  - Pain Consultants of San Diego, La Mesa, California
  - California Orthopedics & Spine, Larkspur, California
  - Remedy Pain Solutions, Inc., Marina del Rey, California
  - Newport Beach Headache & Pain, Newport Beach, California
  - Pain Consultants of San Diego- Poway, Poway, California
  - Relieve Pain Center, San Diego, California
  - Paul Kim MD Pain Management, San Diego, California
  - San Diego Comprehensive Pain Management Center, San Diego, California
  - Source Healthcare, Santa Monica, California
  - Evolve Restorative Center, Santa Rosa, California
  - Innovative Pain Treatment Solutions, Temecula, California
  - Intergrated Pain Management Medical Group, Inc., Walnut Creek, California
  - Front Range Pain Medicine, Fort Collins, Colorado
  - The Orthopaedic & Sports Medicine Center, Trumbull, Connecticut
  - International Spine Pain & Performance Center, Washington D.C., District of Columbia
  - Southeast Spine Associates, Fort Lauderdale, Florida
  - Holy Cross Interventional Spine and Pain Medicine, Fort Lauderdale, Florida
  - Jacksonville Spine Center, Jacksonville, Florida
  - Jupiter Interventional Pain Management, Jupiter, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - Lake Nona Medical Arts, Orlando, Florida
  - Southwest Florida Pain Center, Port Charlotte, Florida
  - Florida Pain Management Associates, Sebastian, Florida
  - Tampa Pain Relief Center, Inc., Tampa, Florida
  - The Spine Center of Southeast Georgia, Brunswick, Georgia
  - Georgia Pain and Spine Care, Newnan, Georgia
  - AXIS Spine Center, Coeur d'Alene, Idaho
  - AMITA Health Bolingbrook Pain Management Center, Bolingbrook, Illinois
  - Rush University Medical Center Department of Anesthesiology, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - Pain Management Center of Paducah, KY, Paducah, Kentucky
  - Pain and Wellness, Cambridge, Massachusetts
  - Columbia Interventional Pain Center, Columbia, Missouri
  - Pain Management Associates, Lee's Summit, Missouri
  - Comprehensive and Interventional Pain Management, Henderson, Nevada
  - Advanced Pain Specialists, Reno, Nevada
  - Center for Pain Control at Jasper Ambulatory Surgical Center, Brick, New Jersey
  - Spine Institute of North America, LLC, East Windsor, New Jersey
  - Premier Pain Center, Shrewsbury, New Jersey
  - University Clinical Research Center, Somerset, New Jersey
  - Pain Management at Garden State Medical Center, Whiting, New Jersey
  - Upstate Orthopedics, East Syracuse, New York
  - Ainsworth Institute of Pain Management, New York, New York
  - Cincinnati Comprehensive Pain Center, Cincinnati, Ohio
  - Dayton Outpatient Center, Dayton, Ohio
  - Summit Medical Center, Edmond, Oklahoma
  - Performance Spine & Sports Physicians, PC, East Norriton, Pennsylvania
  - Center for Interventional Pain & Spine, Exton, Pennsylvania
  - SC Pain and Spine, Murrells Inlet, South Carolina
  - North Lake Pain Consultants, Conroe, Texas
  - Performance Pain and Sports Medicine, Houston, Texas
  - Fondren Orthopedic Group, LLC, Kingwood, Texas
  - Advanced Spine and Pain Center, San Antonio, Texas
  - Precision Spine Care, Tyler, Texas
  - Southwest Spine and Pain, St. George, Utah
  - The Spine and Nerve Center of Saint Francis Hospital, Charleston, West Virginia
  - Advanced Pain Management, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Superion® Indirect Decompression System (IDS)
Started | 1674
Completed | 1594
Not Completed | 80

BASELINE CHARACTERISTICS:
Population: Data as available for study participants is reported.
Arm/Group | Superion® Indirect Decompression System (IDS)
Number analyzed (Participants) | 1601
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data was missing for 5 participants. Data as available for study participants is reported.
  years
    number analyzed (Participants) | 1596
    (all) | 73.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 874
  Male | 727
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline Pain Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Pain score was collected on a scale of 0 -100 (VAS Scale) where 0 is no pain and 100 is worst pain possible. Population: Data is missing for 169 participants. Data as available for study participants is reported.
  units on a scale
    number analyzed (Participants) | 1432
    (all) | 68.6 (26.1)

OUTCOME MEASURES:

1. Primary Outcome: Vertiflex® Patient Satisfaction Survey
Description: Percentage of patients reporting satisfied or somewhat satisfied with treatment during study follow up was calculated.
  Patients chose one of the following options to describe their overall satisfaction with their treatment (1) Satisfied (2) Somewhat Satisfied (3) Somewhat Dissatisfied (4) Dissatisfied. The percentage of patients who reported (1) Satisfied or (2) Somewhat satisfied were included and calculated in the analysis. Maximum is 100% of patients reported being satisfied and minimum is 0%.
Time Frame: 3 Week Follow-Up Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Superion® Indirect Decompression System (IDS)
Number analyzed (Participants) | 1311
Participants | 1147

2. Primary Outcome: Vertiflex® Patient Satisfaction Survey
Description: as for outcome 1
Time Frame: 6 Month Follow-Up Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Superion® Indirect Decompression System (IDS)
Number analyzed (Participants) | 980
Participants | 806

3. Primary Outcome: Vertiflex® Patient Satisfaction Survey
Description: as for outcome 1
Time Frame: 12 Month Follow-Up Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Superion® Indirect Decompression System (IDS)
Number analyzed (Participants) | 763
Participants | 630

ADVERSE EVENTS:
Time Frame: Serious Adverse events (device or procedure related) up to 1 year follow up were only collected. Other adverse events not collected.
Description: Serious Adverse events (device or procedure related) up to 1 year follow up were only collected. Other adverse events not collected.
Arm/Group | Superion® Indirect Decompression System (IDS)
All-Cause Mortality (participants affected / at risk) | 1/1674
Serious Adverse Events (participants affected / at risk) | 5/1674
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Superion® Indirect Decompression System (IDS) (N=1674)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atelectasis (Post-Op) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04087811/Prot_000.pdf